CLINICAL TRIAL: NCT06529679
Title: Mi-SPA: Michigan Split-belt Adaptation Paradigm to Improve Knee Loading After Anterior Cruciate Ligament Reconstruction (Aim 2)
Brief Title: Michigan Split-belt Treadmill Training Program to Improve Acute Knee Biomechanics After ACL Reconstruction
Acronym: Mi-SPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Riann Palmieri-Smith, Professor School of Kinesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00221406_Aim2; 1R21AR082643 (NIH)
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: ACL; ACL Injury
Keywords: Biomechanics; Knee loading; Split-belt; Asymmetric Walking
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Stance Training (Experimental): This study arm will complete both a 20-minute split-belt & tied-belt session. During the split-belt session, the ACL limb will walk at a faster speed (150-170% of 1.1 m/s) than the non-ACL limb (1.1 m/s). During the tied-belt session both limbs will walk at the same speed which will be set to match the faster speed of the ACL leg from the split-belt training day.
  Interventions: Behavioral: Split-belt Training; Behavioral: Tied-Belt Training
- Mid-Stance Training (Experimental): This study arm will complete both a 20-minute split-belt & tied-belt session. During the split-belt session, the ACL limb will walk at a slower speed (30-50% of 1.1 m/s) than the non-ACL limb (1.1 m/s). During the tied-belt session both limbs will walk at the same speed which will be set to match the slower speed of the ACL leg from the split-belt training day.
  Interventions: Behavioral: Split-belt Training; Behavioral: Tied-Belt Training

INTERVENTIONS:
Behavioral: Split-belt Training — Walking on a split-belt treadmill in which the speed of one belt will be different (move faster or slower) than the speed of the other belt.
Behavioral: Tied-Belt Training — Walking on a split-belt treadmill in which the speed of both belts is the same.

SUMMARY:
The goal of this study is to determine short-term adaptations (aftereffects) in knee loading after a 20-minute split-belt treadmill training session in patients with ACL reconstruction.

Our main question for this aim are:

1. Are training-mediated aftereffects in the knee joint moment greater for tied-belt walking or split-belt walking?
2. Are training-mediated aftereffects in the knee joint moment different between subjects who train early stance knee loading versus subjects who train mid-stance knee loading?

DETAILED DESCRIPTION:
Knee and limb underloading are ubiquitous after anterior cruciate ligament (ACL) reconstruction and fails to resolve with the standard of care rehabilitation. This underloading behavior is clinically concerning and considered maladaptive, as it affects patient function, has been linked to risk for re-injury, and appears to be a precursor for post-traumatic knee osteoarthritis that affects upwards of 50% of patients who undergo an ACL reconstruction.

Split-belt treadmill training is a gait retraining approach where treadmill belt speeds are decoupled (i.e., one belt is set to move at a faster or slower speed than the other belt) during walking. Split-belt training is based on well-established motor learning principles, such as error-based learning and variability of practice which can lead to locomotor adaptations. In healthy individuals, split-belt treadmill walking significantly increases knee moment impulses in the limb on the slow belt than on the fast belt during the braking and propulsive phases of gait. Split-belt treadmill training has also shown promise in individuals with neurological deficits, resulting in significant improvements in gait biomechanics after training.

The aim of this project is to determine short-term adaptations (aftereffects) in knee loading after a 20-minute split-belt treadmill training session in individuals with anterior cruciate ligament (ACL) reconstruction. Individuals ~6-10 months after ACL reconstruction will be randomly assigned to 1 of 2 groups and each group will complete a split-belt and tied-belt session. One group will train the early stance knee moment with split-belt walking, while the other group will train the mid-stance knee moment with split-belt walking. Both groups will also complete a tied-belt session. Bilateral knee loading will be quantified using peak knee moments before training (10 min), during training (20 min), and after training (10 min). The investigators hypothesize that the training-mediated aftereffects (i.e., loading after training) will be significantly higher in the split-belt condition than in the tied-belt control condition. The investigators also hypothesize that early stance split-belt training will lead to training-mediated aftereffects for the early stance moment only, while mid-stance training will only result in aftereffects for the mid-stance knee moment.

ELIGIBILITY:
Inclusion Criteria:

* aged 14-45 years
* suffered an acute, complete ACL rupture as confirmed by MRI and physical exam
* have undergone ACL reconstruction w autograft within the past 10 months
* willingness to participate in testing and follow-up as outlined in the protocol
* English-speaking

Exclusion Criteria:

* inability to provide written informed consent
* female subjects who are pregnant or are planning to become pregnant (self-reported)
* previous ACL injury
* previous surgery to either knee
* bony fracture accompanying ACL injury
* patients who experienced a knee dislocation
* patients who had their ACL reconstructed with an allograft
* patients who underwent a multi-ligamentous and/or staged ACL reconstruction

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
ACL Limb Sagittal Plane Knee Joint Moment | Before (10min), during (20min), & after training (10min)
  Peak sagittal plane knee moment recorded from the ACL limb during walking gait

OTHER OUTCOMES:
Non-ACL Limb Sagittal Plane Knee Joint Moment | Before (10min), during (20min), & after training (10min)
  Peak sagittal plane knee moment recorded from the Non-ACL limb during walking gait
ACL Limb Vertical Ground Reaction Force | Before (10min), during (20min), & after training (10min)
  Peak vertical ground recorded from the ACL limb during walking gait
Non-ACL Limb Vertical Ground Reaction Force | Before (10min), during (20min), & after training (10min)
  Peak vertical ground recorded from the Non-ACL limb during walking gait
ACL Limb Internal Knee Joint Reaction Force | Before (10min), during (20min), & after training (10min)
  Internal knee joint reaction force for the ACL limb estimated using musculoskeletal modeling
Non-ACL Limb Internal Knee Joint Reaction Force | Before (10min), during (20min), & after training (10min)
  Internal knee joint reaction force for the Non-ACL limb estimated using musculoskeletal modeling

CONTACTS AND LOCATIONS:
Overall Officials: Riann M Palmieri-Smith, PhD, ATC, Principal Investigator — University of Michigan; Chandramouli Krishnan, PT, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made publicly available via Deep Blue Data which is managed by the University of Michigan.
Supporting Information: Study Protocol, ICF
Time Frame: We will strive to release data to the repository as rapidly as it is possible to analyze experiments and publish results. Data used in publications will be released at the time of publication.